CLINICAL TRIAL: NCT05095415
Title: The Effect of an Occupational Therapy Pre-operative Education Consult on Patient Outcomes in the Orthopedic Hand Setting: A Prospective Randomized Block Study
Brief Title: Occupational Therapy Pre-operative Education in the Orthopedic Hand Setting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator has left the institution (graduated)
Sponsor: Methodist University, North Carolina (Other)
Collaborators: Cape Fear Orthopedics & Sports Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MethodistUNC
Record Dates: First submitted 2021-09-21; First posted 2021-10-27 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2021-10

CONDITIONS: Flexor Tendon Rupture; Thumb Osteoarthritis; Distal Radius Fracture
Keywords: Occupational Therapy; Pre-operative Education; Upper Extremity
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the experimental or control group in accordance with their diagnosis specific block. This will be continued until there is at least 5 participants in each diagnosis block.
Who Masked: Participant
Masking Description: Participants will be masked to the knowledge of if they are receiving the typical pre-operative care or an additional individualized occupational therapy consult.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Typical Pre-operative Experience (Active Comparator): Participants will be be placed in appropriate subgroups based upon their diagnosis and surgical intervention. Subgroups include: CMC Arthroplasty, ORIF of the Distal Radius, and Flexor/Extensor Tendon Repairs.
  Interventions: Other: Typical Pre-Operative Education
- Occupational Therapy Consult Experience (Experimental): Participants will be be placed in appropriate subgroups based upon their diagnosis and surgical intervention. Subgroups include: CMC Arthroplasty, ORIF of the Distal Radius, and Flexor/Extensor Tendon Repairs.
  Interventions: Other: Occupational Therapy Pre-operative Consult

INTERVENTIONS:
Other: Occupational Therapy Pre-operative Consult — Preoperative education will be given by the treating orthopedic surgeon first and will then be followed by a consult with a final semester, occupational therapy student. The pre-operative education will include the importance of attending therapy, what to expect at therapy, typical duration of therapy for their specific diagnosis, and address any questions of ther participant. Participants will be given educational materials and access to education videos to watch if they so choose.
  Arms: Occupational Therapy Consult Experience
Other: Typical Pre-Operative Education — Participants will receive all preoperative education from their orthopedic surgeon and will not be spoken to directly about the therapeutic process until their first scheduled therapy appointment.
  Arms: Typical Pre-operative Experience

SUMMARY:
This will be a prospective randomized control trial with a blocking method to determine the effect of an occupational therapy focused pre-operative education on 3 pre-determined diagnosis: Carpometacarpal (CMC) Arthroplasty, Distal radius fracture requiring open reduction internal fixation (ORIF) and tendon repairs of the hand. Possible participants will be recruited through Cape Fear Orthopedics & Sports Medicine and receiving care from an orthopedic surgeon & hand specialist. Researchers hypothesize that those who receive the occupational therapy consult will demonstrate improved adherence with occupational therapy appointments, improved patient perceived function, and overall improved experiences with the pre-operative patient experience.

DETAILED DESCRIPTION:
Participants will be identified by orthopedic surgeon. Once informed consent is obtained participants will subsequently be randomly assigned to the control or experimental block associated with their diagnosis. Patients will be randomly assigned within their diagnosis block through random number generation in Microsoft Excel. Participants randomly assigned to the control group will receive the current & typical educational information provided by their orthopedic surgeon. Participants randomly assigned to the experimental group will receive an additional occupational therapy (OT) focused pre-operation education consultation provided by a third year occupational therapy student under the supervision of an orthopedic surgeon & Occupational Therapist & Certified Hand Therapist. The additional OT pre-operative consult will be included during participants scheduled pre-operative appointment. Specific pre-op appointments are only conducted when patients have not been seen by a provider within 4-weeks of their surgical date. If surgery is scheduled within 4-weeks of the patients last encounter with a provider an additional pre-op visit is not required. Since two of the three pre-determined diagnosis of interest are typically associated with trauma, participants may receive their OT consult at their first encounter with the orthopedic surgeon which is also considered their pre-op visit.

The OT consult provided to the individuals assigned to the experimental group will consist of a one-on-one interaction with a third year occupational therapy doctorate (OTD) student providing diagnosis specific educational materials inclusive of what to expect after surgery, the importance of attending therapy as recommended by the orthopedic surgeon and how to accurately complete the Upper Extremity Functional Index (UEFI). Outcomes of this research will include UEFI scores at therapeutic evaluation, after 10 visits and upon discharge, completion of a post operative survey via question pro utilizing a Visual Analog Scale (VAS) at the initial therapeutic encounter, and patient compliance with attending therapy as documented by therapy visit attendance. A semi-structured interview will be completed at patient discharge from therapy to determine areas of possible improvement and further research.

Individuals randomly assigned to the control group will participate in the typical pre-operative experience provided by the orthopedic surgeon. Control group participants will not be made aware of experimental group participants experiences. Participants in the control group will be informed that researchers are interested in the pre-operative patient experiences at Cape Fear Orthopedics & Sports Medicine and their participation in the study and honest responses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Distal Radius Fracture, requiring open reduction internal fixation
* Clinical diagnosis of flexor tendon of the hand laceration
* Clinical diagnosis of CMC arthritis, electing to undergo CMC arthroplasty
* Receiving care from Cape Fear Orthopedics & Sports Medicine
* English Speaking

Exclusion Criteria:

* Less than 18 years old
* Previously sustained one of the inclusion criteria diagnoses
* Elect not to receive therapeutic services at Cape Fear Orthopedics & Sports Medicine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Patient appointment attendance | Through completion of therapy, up to one year.
  Patient adherence to scheduled occupational therapy visits
Upper Extremity Functional Index | Date of first attended postoperative therapeutic appointment, up to 15 days following surgery
  Patient reported outcome measure used to assess the functional impairment individuals with musculoskeletal upper limb dysfunction
Upper Extremity Functional Index | Date of 10th attended postoperative therapeutic appointment, up to 30 days following initial therapeutic evaluation
  Patient reported outcome measure used to assess the functional impairment individuals with musculoskeletal upper limb dysfunction
Upper Extremity Functional Index | Upon discharge from therapeutic services, up to one year
  Patient reported outcome measure used to assess the functional impairment individuals with musculoskeletal upper limb dysfunction

SECONDARY OUTCOMES:
QuestionPro Post-Operative Survey using Visual Analogue Scale (VAS) | Date of first attended postoperative therapeutic appointment, up to 15 days following surgery
  Patient reported outcome analyzing patient pre-operative experiences. VAS is linear scale where participants visually mark the line corresponding to their preoperative experience. Patients are blinded to the numerical value associated to their answer to decrease biases. VAS is ten point linear scale where 1 represents the negative anchor and 10 represents the positive, preferred response. Questions address anxiety, understanding, and overall preoperative experience.

IPD SHARING:
Plan to Share IPD: No